CLINICAL TRIAL: NCT03261908
Title: A Pharmacogenomics Study of Simvastatin-Induced Adverse Drug Reaction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy，M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2016[1237]
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Simvastatin Adverse Reaction; Pharmacogenomics; Accurate Medication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wild genotype: Through next generation sequencing, distinguish wild genotype of simvastatin
  Interventions: Genetic: detection of genotype
- mutant genotype: Through next generation sequencing, distinguish mutant genotype of simvastatin
  Interventions: Genetic: detection of genotype

INTERVENTIONS:
Genetic: detection of genotype — detection of genotype by next generation sequencing

SUMMARY:
Adverse reactions of simvastatin are mostly slight and transient, however, the incidence of simvastatin-induced hepatic impairment and myopathy are obviously higher in Chinese population than other racial groups. There is still lack of research data in Chinese. In this study, we will investigate whether there are specific genotypes which may predict the incidence of simvastatin-induced hepatic impairment and myopathy in Chinese so as to provide a basis for developing guidelines on precise medication in simvastatin therapy apply to Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking simvastatin therapy
* Signed informed consent.

Exclusion Criteria:

* Patients not taking simvastatin therapy
* Intolerance or unwillingness to blood sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Patients:In accordance with anti-hyperlipemia indications of simvastatin
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of hepatic impairment | At 2 years
Incidence of myopathy | At 2 years

SECONDARY OUTCOMES:
Genotype detected by next generation sequencing | pre-dose of simvastatin(Baseline)
  Collect blood specimen before simvastatin administration, then detect genotype of simvastatin by next generation sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China